CLINICAL TRIAL: NCT06024889
Title: Acute Effects of Furosemide on Hemodynamics and Pulmonary Congestion in Acute Decompensated Heart Failure.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johannes Grand (Other)
Responsible Party: Sponsor-Investigator, Johannes Grand, Principal Investigator, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-23029822
Record Dates: First submitted 2023-08-23; First posted 2023-09-06 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Furosemide (Experimental): 80 mg of furosemide is administered IV
  Interventions: Drug: Furosemide Injection

INTERVENTIONS:
Drug: Furosemide Injection — Intravenous administration of 80 mg furosemide is followed by assessing blood pressure, peripheral oxygen saturation, pulmonary fluid content by ReDS*, and ultrasound examination of heart and lungs, including assessment of filling pressures with doppler and strain analysis. These measurements are repeated at multiple time points until 6 hours have elapsed.

SUMMARY:
Intravenous (IV) loop diuretics have been a key component in treating pulmonary edema since the 1960s and has a Class 1 recommendation in the 2021 guidelines for acute heart failure. However, no randomized clinical trials have investigated loop diuretics versus other interventions for acute heart failure, and clinical knowledge of the hemodynamic effects of furosemide is based in studies from the 1970s. In this study, we aim to assess the acute effect of furosemide on cardiac filling pressures and pulmonary congestion.

Hypothesis:

Administration of furosemide induces a hyperacute (within 30 minutes) lowering of cardiac filling pressures and pulmonary congestion before significant diuresis occurs.

Design:

A prospective, interventional study including 20 patients admitted due to a clinical diagnosis of acute heart failure with pulmonary congestion.

Intervention:

80 mg of furosemide is administered IV. Measurements include blood pressure, peripheral oxygen saturation, pulmonary fluid content by ReDS*, ultrasound examination of heart and lungs, and assessment of cardiac filling pressures with doppler and strain analysis. Measurements are repeated at several time points until 6 hours have passed.

DETAILED DESCRIPTION:
Prospective observational study of the acute and subacute effects of furosemide in patients with acute heart failure.

After inclusion, 80 mg of furosemide is administered IV.

Measurements include blood pressure, peripheral oxygen saturation, pulmonary fluid content, ultrasound examination of heart and lungs, and assessment of cardiac filling pressures with doppler and strain analysis. Measurements are repeated at several time points until 6 hours have passed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Clinical diagnosis of acute heart failure requiring hospitalization
3. Systolic blood pressure ≥100 mmHg
4. Oxygen saturation <94% or need of oxygen
5. Confirmed pulmonary congestion on x-ray or ReDS

Exclusion Criteria:

1. More than 40 mg iv furosemide within the last three hours before randomization, including prehospital administration
2. Ongoing ventricular taky- or brady-arrythmias or supraventricular arrhythmias with HR > 180 or < 40 bpm.
3. Known chronic obstructive lung disease
4. Pacemaker or ICD on the right side
5. Congenital heart malformations or intra-thoracic mass that would affect the right lung anatomy (e.g. dextrocardia, lung carcinoma)
6. Wounds, burns, healing tissue, skin infection or recent skin graft or flap where the sensors should be attached to the skin
7. Height less than 155 cm or higher than 200 cm
8. BMI of less than 18 or more than 38

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Pulmonary fluid content | From the time 0 to 30 minutes
  Remote dielectric sensing (ReDS) is a non-invasive electromagnetic-based tool that measures absolute lung fluid content and gives the fluid content in a proportional value ranging from 0-100 percent. 20-35% represent normal values.
  The primary outcome will be change in pulmonary fluid content after administration of furosemide

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Grand, Principal Investigator — Department of Cardiology
Locations (1):
- Amager-Hvidovre Hospital, Copenhagen, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Caidi NO, Lukoschewitz JD, Nielsen OW, Hove J, Seven E, Dixen U, Grund F, Petersen M, Foss NB, Grand J. The acute effects of furosemide in acute heart failure assessed by remote dielectric sensing. A protocol. Dan Med J. 2024 Jun 12;71(7):A11230697. doi: 10.61409/A11230697. PMID 38903022